CLINICAL TRIAL: NCT05006846
Title: Technology Improving Success of Medication-Assisted Treatment in Primary Care - Phase 1
Brief Title: Technology for MAT in Primary Care - Phase 1
Status: Completed | Type: Observational
Sponsor: Q2i, LLC (Industry)
Collaborators: University of California, Los Angeles (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-001938; 4R42DA050398-02 (NIH)
Record Dates: First submitted 2021-08-12; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Opioid-use Disorder
Keywords: Opioid use disorder; Primary care; Technological solutions; Medication for opioid use disorder; mHealth
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Primary care physicians (PCPs) and their patients used the intervention (OARS) for 4 weeks. They completed 2 interviews to obtain their feedback on the acceptability and feasibility of using OARS in a primary care setting. Data for this cohort was collected between February 18, 2020, to May 25, 2020.
  Interventions: Other: Opioid Addiction Recovery Support Software Platform
- Cohort 2: Primary care physicians (PCPs) and their patients used the intervention (OARS) for 4 weeks. They completed 2 interviews to obtain their feedback on the acceptability and feasibility of using OARS in a primary care setting. Data for this cohort was collected between July 17, 2020, to August 31, 2020.
  Interventions: Other: Opioid Addiction Recovery Support Software Platform

INTERVENTIONS:
Other: Opioid Addiction Recovery Support Software Platform — OARS (Opioid Addiction Recovery Support) is used by providers of MAT programs to improve insight into a patient's recovery progress while promoting ownership and adherence to treatment plans. OARS also provides extensive tools to support patients with recovery from Opioid Use Disorder.
  Other Names: OARS

SUMMARY:
With over 72,000 overdose deaths in 2017, of which 47,600 are attributable to opioid overdose, the opioid epidemic has become North America's most widespread behavioral public health problem. Medication-assisted treatment (MAT) for opioid use disorder (OUD) is highly efficacious. The Opioid Addiction Recovery Support (OARS), comprised of a healthcare team portal connected to a patient mobile application, provides opioid-related education, promotes connectedness with clinicians, and tracks MAT treatment progress. This study will conduct interviews with patients that will inform optimal design of OARS, assess the efficacy of OARS in improving MAT outcomes in primary care settings, and evaluate the sustainability and return on investment.

It joins an outstanding scientific team at University of California, Los Angeles and a small business that has developed, Opioid Addiction Recovery Support (OARS) -- a software platform that by integrating with the Electronic Health Record (EHR) improves clinical management of patients by primary care providers (PCPs) treating patients with OUD using MAT. OARS platform uses a dashboard to show the real-time measurement of patient achievements in recovery. It provides opportunities for patients to interact with their PCPs, allowing for better connection to and support from their PCPs. OARS platform features artificial intelligence to analyze information from the EHR and from patients to provide a relapse risk assessment for patients receiving MAT for OUD, an innovation that sets OARS apart from other software solutions. The goal of Phase 1 was to modify the OARS platform for use in primary care settings by conducting interviews with Primary Care Physicians (PCPs) (N=20) and their patients with OUD (N=40) in primary care settings to collect data on feasibility and acceptability of engaging with OARS to inform the user-centered design of OARS.

ELIGIBILITY:
Inclusion Criteria:

* For PCPs: (1) physician, nurse practitioner, or physician's assistant in any area within primary care; (2) in possession of valid DATA-2000 waiver; (3) currently treating more than two patients with OUD using oral buprenorphine-naloxone product; (4) willing to distribute study materials to their patients describing the research and providing options for their participation.
* For patient participants: (1) diagnosed and treated using MAT within primary care setting (i.e., family medicine, internal medicine, adolescent medicine, pediatrics, obstetrics/gynecology, geriatrics, infectious diseases, emergency department, non-cancer pain management

Exclusion Criteria:

* For PCPs: (1) specialization outside primary care (e.g., psychiatry, neurology, etc) or provider works in specialized setting (e.g., addiction treatment programs; mental health clinic); (2) not treating patients with OUD with oral buprenorphine-naloxone product (e.g., long-acting naltrexone or buprenorphine injections); (3) Individual interviews with physicians and their patients to discuss initially barriers and challenges to MAT for patients with OUD seen in primary care settings.
* For patient participants: (1) MAT delivered in specialty care settings (i.e., psychiatry, substance abuse treatment programs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary care providers (PCPs) willing to prescribe buprenorphine-naloxone and willing to allow two of their patients with OUD to participate were recruited through mailed recruitment flyers and by reaching out to individual clinics.
  Patients were recruited through their PCP, with a maximum of two patients per PCPs participating in the study using passive recruitment of patients via email describing the study which is used so that potential patient participants can elect to or not engage in this research project independent of their PCPs decisions. Recruitment materials clarified that patients' decisions regarding research participation did in no way impact patients' clinical care. Patients whose PCPs elected not to participate in this research were also not eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility for primary care providers (PCPs) | From week 1 to week 4.
  Frequency of days of engagement per week and use of interactive features does not reduce over 20%.
Feasibility for patients | From week 1 to week 4.
  Frequency of days of engagement per week and use of interactive features does not reduce over 20%.
Acceptability for PCPs | At week 4.
  No more than 20% of qualitative mentions that describe barriers or dissatisfactions with using OARS platform).
Acceptability for patients | At week 4.
  No more than 20% of qualitative mentions that describe barriers or dissatisfactions with using OARS platform).

SECONDARY OUTCOMES:
System Usability Scale for providers | At week 4.
  The System Usability Scale (SUS) is a tool for measuring the usability, consisting of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree.
System Usability Scale for patients | At week 4.
  The System Usability Scale (SUS) is a tool for measuring the usability, consisting of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Shoptaw, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Behavioral and Addiction Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Further information about the OARS solution available here. — http://q2i.com/oars/